CLINICAL TRIAL: NCT03107117
Title: Computer-Assisted Brief Intervention Protocol for Marijuana Using Juvenile Offenders
Brief Title: Computer-Assisted Brief Intervention
Acronym: JJMISCOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Anthony Spirito, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DA042247
Record Dates: First submitted 2017-03-31; First posted 2017-04-11 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: a computer-assisted adolescent motivational interview plus an online parenting program for substance abuse will be compared to usual care.
Who Masked: Outcomes Assessor
Masking Description: Blind to treatment condition to which subject is assigned
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer counseling (Experimental): a computer-assisted adolescent motivational intervention called e-toke plus an online parenting program - Parenting Wisely
  Interventions: Behavioral: Computer Counseling
- Standard care (Active Comparator): Standard care is typically referral to counseling for substance use
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Computer Counseling — two computer counseling online programs for a teen and a parent
  Arms: Computer counseling
Behavioral: Standard Care — A referral for substance use counseling
  Arms: Standard care

SUMMARY:
Due to the "unmet needs" of substance abuse treatment among court involved but non-incarcerated (CINI) adolescents and their parents, reaching and engaging CINI adolescents in intervention programs addressing marijuana use is important given the significant risk that continued substance use poses for re-arrest and detention. This study will examine the feasibility of implementing one potential model for increasing access to substance use interventions in a juvenile justice setting by using: 1) a computer- assisted intervention addressing marijuana use for adolescents, and 2) a computer program on strategies to improve management of teens who misuse drugs for parents.

DETAILED DESCRIPTION:
Four out of five youth in the juvenile justice system show evidence of being under the influence during their offenses, and over half test positive for substances at the time of their arrest. Further, 92% of arrested juveniles who tested positive for drugs tested positive for marijuana. Although some treatment programs for juvenile offenders exist, most have focused on detained and incarcerated juveniles, who only represent one third of arrested youth. As a result, little is known about how to improve the continuum of care for the remaining two-thirds of this population, which consists of court involved but non-incarcerated youth (CINI). Court recommendations and referrals for CINI have mostly relied on outside community-based services, thus decreasing the likelihood CINI youth and their families will take the additional steps to seek intervention. Given that motivational interventions (MI) are brief, relatively easy to implement and have a greater reach than typical substance use treatment programs, researchers have recently directed their focus to interactive, computer-delivered MI protocols to further increase their reach as well as facilitate their implementation. Online interventions can be delivered at a lower cost, with less demand on staff time for training, and increased protocol fidelity, portability, and ease of use. While counselor-delivered MIs for adolescent substance use have been tested fairly widely, only a few studies have been published on the efficacy of computer-assisted MIs. Further, little research has focused on the efficacy of such interventions with marijuana using adolescents in general, and more specifically with CINI adolescents. In addition, combining such interventions for adolescents with brief parenting interventions is important but yet rarely implemented. Therefore, this application proposes to examine the feasibility and acceptability of integrating a computer-assisted,, brief intervention protocol into the juvenile intake procedures at the Rhode Island Family Court (RIFC) for marijuana using adolescents and their parents. Following an open trial of the brief protocol, , 80 adolescents who screen positive for marijuana use at juvenile intake will be recruited from the RIFC and randomly assigned to one of two conditions: 1) a computer-assisted adolescent MI plus an online parenting program ; or 2) usual care. Outcomes will be examined at 3 and 6-month follow-ups. This small trial will provide some initial evidence regarding utility of this protocol with CINI youth and whether a larger, fully powered trial is indicated in the future.

ELIGIBILITY:
Inclusion Criteria:

* teen age 14 to 17, inclusive, living at home with at least one parent/guardian
* teen report of history of marijuana use and a positive brief screen during intake procedures * parental consent/ child assent; and, 4) one parent willing to participate in intervention

Exclusion Criteria:

* developmental delay
* teen or parents are not able to adequately speak and understand English or Spanish.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Time Line Follow Back Interview (TLFB) | 90 days
  The Timeline Follow-back Interview is a widely used research tool with good reliability and validity for various groups of individuals. Marijuana and alcohol consumption information is collected using a calendar format with temporal cues (e.g., holidays) to assist in recall of days when marijuana and alcohol were used. Data from the TLFB will be summarized to yield the total number of marijuana and alcohol use days.

SECONDARY OUTCOMES:
Marijuana and alcohol problems | 90 days
  Marijuana and alcohol use problems will be assessed using items from the Add Health longitudinal study on symptoms of abuse and dependence including problems at school, home; physical fights; and physical symptoms such as vomiting and "hang over."

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Spirito, PhD, Principal Investigator — Brown University
Locations (1):
- Rhode Island Family Court, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Analysis files will be constructed from the stored electronic data and will be stripped of identifying information with the Safe Harbor method. Specifically, youth and their parents will be identified with a family identifier and person identifier number that is randomly generated and not related to any element of their personal identifying information. No names, addresses, telephone numbers, fax numbers, email addresses, social security numbers, medical records, etc. will be retained. Dates will contain only year and a randomly generated day-of-the-year. We will only share it with external investigators when a data use agreement (DUA) is executed between the Brown University and the requester's institution. The DUA will specify the requested data elements (each of which must be justified), the specific research question, the timeline for the project, and schedule for data destruction. The data will be made available on April 1, 2021 by the PI

DOCUMENTS (1):
  • Informed Consent Form (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT03107117/ICF_000.pdf